CLINICAL TRIAL: NCT07310277
Title: Expanded Access to ABBV-706
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C25-216
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ABBV-706 — Intravenous (IV) Infusion

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to ABBV-706 prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=C25-216